CLINICAL TRIAL: NCT02501005
Title: Preventive aBlation of vEntricular tachycaRdia in Patients With myocardiaL INfarction
Acronym: BERLIN VT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to futility
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP028
Record Dates: First submitted 2015-07-06; First posted 2015-07-17 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group 1 (TG1) (Experimental): Prophylactic VT ablation prior to ICD implantation
  Interventions: Procedure: VT ablation
- Treatment Group 2 (TG2) (Other): ICD implantation and best medical care until the third appropriate ICD shock occurs and catheter ablation thereafter
  Interventions: Procedure: VT ablation

INTERVENTIONS:
Procedure: VT ablation — Catheter ablation of ventricular tachycardia

SUMMARY:
The BERLIN VT study is designed to evaluate the impact of prophylactic ventricular tachycardia (VT) ablation on all-cause mortality and unplanned hospital admission for congestive heart failure or symptomatic ventricular tachycardia/ventricular fibrillation (VF) when compared to VT ablation after the third appropriate implantable cardioverter-defibrillator (ICD) shock.

ELIGIBILITY:
Inclusion Criteria:

1. History of remote myocardial infarction
2. Left ventricular ejection fraction ≥ 30 to ≤ 50 % as estimated by cardiac MRI, 3D-echocardiography or via ventriculography within 30 days before enrollment
3. Documentation of sustained ventricular tachycardia (VT) by any kind of Electrocardiography (ECG) including 12 lead ECG, holter ECG, rhythm strip, event monitoring, event recorder or pacemaker within 30 days before enrollment
4. Implantable cardioverter-defibrillator (ICD) indication for secondary prevention
5. Patients who are planned to be implanted with BIOTRONIK ICDs (single, dual, triple chamber or DX device)
6. Patient has provided written informed consent
7. Patient accepts activation of Home Monitoring®

Exclusion Criteria:

1. Age < 18 years or > 80 years
2. Known arterial or venous thrombosis
3. Class IV New York Heart Association (NYHA) heart failure
4. Valvular heart disease or mechanical heart valve precluding access to the left ventricle
5. Acute myocardial reinfarction or acute coronary syndrome
6. Cardiac surgery involving cardiotomy within the past 2 months
7. Patients requiring chronic renal dialysis
8. Thrombocytopenia or coagulopathy
9. Incessant VT or electrical storm
10. Bundle branch reentry tachycardia as the presenting VT
11. Pre-existing implantable cardioverter-defibrillator (ICD)
12. Pregnancy or breast feeding women
13. Acute illness or active systemic infection
14. Other disease process likely to limit survival to less than 12 months
15. Significant medical problem that in the opinion of the principal investigator would preclude enrollment in the study
16. Unwillingness to participate or lack of availability for follow-up
17. Participation in another interventional clinical investigation during the course of the study, i.e. the participation in a non-interventional clinical investigation is allowed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Time to first event comprising all-cause mortality, unplanned hospital admission for congestive heart failure and unplanned hospital admission for symptomatic ventricular tachycardia (VT)/ ventricular fibrillation (VF) | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.

SECONDARY OUTCOMES:
Time to first sustained ventricular tachycardia (VT)/ ventricular fibrillation (VF) | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months..
Time to first appropriate implantable cardioverter-defibrillator (ICD) therapy | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Time to first inappropriate implantable cardioverter-defibrillator (ICD) therapy | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Time to all-cause mortality | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Time to cardiac mortality | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Time to first unplanned all-cause hospitalization | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Time to first unplanned cardiac hospitalization | From randomization until official study end or drop-out, patients will be followed and assessed for primary endpoint events and Time-to-Event Outcome Measures for an expected average of 30 months.
Changes in quality of life / mental | 12 months
  This endpoint compares the changes in the mental component score of the Short Form-36 (SF-36) questionnaire from enrollment to the 12-months follow-up. Additionally, descriptive statistics is calculated: absolute scores at enrollment, 3-month follow-up, and 12-month follow-up, short-term changes in scores from enrollment to the 3-month follow-up.
Changes in quality of life / physical | 12 months
  This endpoint compares the changes in the physical component score of the Short Form-36 (SF-36) questionnaire from enrollment to the 12-months follow-up. Additionally, descriptive statistics is calculated: absolute scores at enrollment, 3-month follow-up, and 12-month follow-up, short-term changes in scores from enrollment to the 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof., Principal Investigator — Asklepios Klinik St. Georg, Hamburg (Germany); Stephan Willems, Prof., Study Chair — Universitäres Herzzentrum, Hamburg (Germany)
Locations (5):
- Germany (5):
  - Universitätsklinikum Köln, Cologne
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Klinikum der Universität München, München

REFERENCES:
- [Background] Tilz RR, Kuck KH, Kaab S, Wegscheider K, Thiem A, Wenzel B, Willems S, Steven D. Rationale and design of BERLIN VT study: a multicenter randomised trial comparing preventive versus deferred ablation of ventricular tachycardia. BMJ Open. 2019 May 9;9(5):e022910. doi: 10.1136/bmjopen-2018-022910. PMID 31072848
- [Derived] Willems S, Tilz RR, Steven D, Kaab S, Wegscheider K, Geller L, Meyer C, Heeger CH, Metzner A, Sinner MF, Schluter M, Nordbeck P, Eckardt L, Bogossian H, Sultan A, Wenzel B, Kuck KH; BERLIN VT Investigators. Preventive or Deferred Ablation of Ventricular Tachycardia in Patients With Ischemic Cardiomyopathy and Implantable Defibrillator (BERLIN VT): A Multicenter Randomized Trial. Circulation. 2020 Mar 31;141(13):1057-1067. doi: 10.1161/CIRCULATIONAHA.119.043400. Epub 2020 Jan 31. PMID 32000514
- See also: Design Paper — https://www.ncbi.nlm.nih.gov/pubmed/31072848